CLINICAL TRIAL: NCT00937768
Title: Phase II Trial of Temporary Androgen Deprivation Therapy in High Risk Prostate Cancer Following Radical Prostatectomy
Brief Title: Leuprolide Acetate or Goserelin Acetate Compared With Observation in Treating Patients With High-Risk Prostate Cancer Who Have Undergone Radical Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC0852; NCI-2009-01147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08-001519; MC0852 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2018-12

CONDITIONS: Prostate Adenocarcinoma; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (antihormone therapy) (Experimental): Patients receive leuprolide acetate IM on day 1 OR goserelin acetate SC on day 1. Courses repeat every 3 months for 9 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment
- Arm B (no antihormone therapy) (No Intervention): Patients undergo observation every 3 months for 9 months.

INTERVENTIONS:
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
  Arms: Arm A (antihormone therapy)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm A (antihormone therapy)
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
  Arms: Arm A (antihormone therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm A (antihormone therapy)

SUMMARY:
This randomized phase II trial studies the side effects and how well giving leuprolide acetate or goserelin acetate works compared to observation in treating patients with high-risk prostate cancer who have undergone radical prostatectomy. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as goserelin acetate and leuprolide acetate, may lessen the amount of androgens made by the body and thus control prostate cancer growth. Many times, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. However, in some prostate cancers there is a chance that tumors can re-grow despite surgery based on certain high risk features.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the difference in the biochemical progression-free survival rate (bPFS) at 2-years between immediate androgen deprivation therapy (ADT) for nine months in high risk prostate cancer patients following radical prostatectomy and a similar high risk patient population followed without initiation of immediate ADT treatment.

SECONDARY OBJECTIVES:

I. To determine the difference in bPFS, prostate cancer specific survival, and overall survival between immediate ADT for nine months and observation for high risk prostate cancer patients following radical prostatectomy.

II. To evaluate the toxicity profile and quality of life (QOL) measured by Functional Assessment of Cancer Therapy-Prostate (FACT-P) and linear analogue self assessment (LASA) between two treatment arms.

TERTIARY OBJECTIVES:

I. To explore if serum and urine biomarker(s) levels at study entry, 9 months, or 24 months in the two treatment arms are correlated with biochemical progression-free survival rate.

II. To explore if > 5 circulating tumor cells (CTCs) or circulating endothelial cells (CECs) following study treatments are associated with biochemical progression-free survival rate.

III. To explore the prognostic and predictive value of tissue based biomarkers in high risk prostate cancer patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive leuprolide acetate intramuscularly (IM) on day 1 OR goserelin acetate subcutaneously (SC) on day 1. Courses repeat every 3 months for 9 months in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo observation every 3 months for 9 months.

After completion of study treatment, patients are followed up every three months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION:
* Informed consent explained and signed prior to any study related procedures
* Patients with any one of the following "high risk" criteria:

  * Clinical or pathological Gleason score 8-10
  * Prostate-specific antigen (PSA) > 20 ng/ml at initial presentation prior to radical prostatectomy
* Willingness to provide mandatory tissue for research purposes
* Willingness to provide mandatory blood for research purposes
* Has no history of androgen deprivation therapy within the past 6 months or has been treated neoadjuvantly up to 6 months prior to radical prostatectomy with the following agents; luteinizing hormone-releasing hormone (LHRH) agonists, anti-androgens, 5 alpha-reductase inhibitors, and peripheral anti-androgens
* REGISTRATION:
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2; or Karnofsky performance of > 60%
* Patients with any one of the following "high risk" criteria:

  * Gleason, prostate specific antigen, seminal vesicle and margin status (GPSM) score >= 10 [GS + 1*(PSA 4-10)+2*(PSA 10.1-20)+3*(PSA > 20)+2*(seminal vesicular or nodal involvement) +2*(margin)](determined post radical prostatectomy)
  * Post prostatectomy seminal vesicle invasion (pT3b) or pT4
  * Two or less microscopic lymph nodal metastasis determined at the time of prostatectomy OR
  * Gleason 4+3 at the time of prostatectomy with margin positivity
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 2 x institutional upper limit of normal (ULN)
* Total bilirubin =< 2 x institutional ULN
* For patients identified as high-risk on the basis of pathological criteria after undergoing radical prostatectomy: interval time for study enrollment after radical prostatectomy will be =< 28 days of the prostatectomy
* For patients identified as high-risk prior to undergoing radical prostatectomy: patients presenting with a high Gleason score (8-10) and/or a PSA > 20 ng/ml are deemed eligible for study participation and study registration as long as the eligibility criteria is reconfirmed post radical prostatectomy; these patient groups may choose to register prior to or after prostatectomy
* Study randomization must occur =< 28 days of radical prostatectomy; all patients consented on the trial, whether consented in the pre-prostatectomy or post-prostatectomy period, will be randomized to study treatments =< 28 days of prostatectomy
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* PRE-REGISTRATION
* Transitional cell, small cell, or squamous cell carcinoma of the prostate; NOTE: patients consented for participation prior to prostatectomy, if detected to have above listed histo-pathologies after prostatectomy will be deemed ineligible and not proceed to study randomization
* History of primary prostate cancer treatment
* Evidence of clinical nodal disease (N1) or grossly evident metastasis at the time of enrollment
* History of bilateral orchiectomy; unilateral orchiectomy with normal range serum testosterone levels will be allowed for enrollment
* Evidence of metastasis on radiographic metastatic workup within a preceding period of 4 months from the time of study entry, including whole body radionuclide bone scan, computed tomography (CT) and/or magnetic resonance (MR) scan of the pelvis and abdomen; otherwise will perform at the time of the baseline tests and result must be normal to continue on study; results of ProstaScint or other radionuclide scans, excluding radionuclide bone scans, will NOT be used to establish metastatic disease if all other studies are negative
* Receiving other experimental drugs =< 4 weeks prior to consenting
* Uncontrolled infection
* History of other cancer, excluding squamous cell and basal cell skin cancers, within the preceding 2 years
* Documented history of human immunodeficiency virus (HIV) positivity or other acquired immunodeficiency disorder, congenital immunodeficiency disorder, or history of organ transplantation
* Unable to follow up every three months for the first year to Mayo Clinic, Rochester for receiving LHRH analogues or study monitoring
* REGISTRATION:
* Uncontrolled infection
* Unable to follow up every three months for the first year to Mayo Clinic, Rochester for receiving LHRH analogues or study monitoring

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Karnes, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen (16) participants were recruited at Mayo Clinic (Rochester) between July 2009 and June 2012.
Pre-assignment Details: This trial was terminated early due to funding issues.
Groups:
- Androgen Deprivation Therapy: Patients receive leuprolide acetate intramuscularly (IM) on day 1 OR goserelin acetate subcutaneously (SC) on day 1.
- No Androgen Deprivation Therapy: Patients undergo observation every 3 months for 9 months.
Period: Overall Study
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8
Not completed — Refused Further Treatment | 3 | 2
Not completed — Disease Progression | 1 | 1
Not completed — Alternate Treatment | 0 | 1
Not completed — No Further Funding | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.6) | 62.8 (7.4) | 62.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Progression-free Survival Rate
Description: Biochemical progression-free survival (BPFS) was defined as the time from randomization to the time of biochemical progression. If a patient dies without a documentation of biochemical progression, the patient will be considered to have had progressed at the time of death.
Time Frame: 2 years
Population: No participants reached the 2 years follow up due to the early termination of the trial.
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Deaths
Description: The number of deaths due to any cause are reported below.
Time Frame: 2 years
Population: Study terminated prematurely due to funding issues. Planned analysis for Overall Survival and Prostate Cancer Specific Survival was not performed due to the nature of the closure. Thus, the number of deaths are reported below.
Measure: Count of Participants; unit: Participants
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events Regardless of Attribution
Description: Percentage of Participants with Grade 3 or Higher Adverse Events regardless of attribution per NCI CTCAE Version 3
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 8 | 8
percentage of patients | 100 | 37.5

4. Secondary Outcome: Average Overall FACT-P Total Score at Baseline, Months 3 and 6
Description: The overall FACT-P Total Score at Baseline and months 3 and 6 mean and standard deviations are reported below. The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain, as well as a global quality of life score which is the sum of all 5 domain scores and ranges from 0 to 156 where higher scores represent better quality of life.
Time Frame: Baseline and months 3 and 6
Population: Patients who completed the FACT-P and had FACT-P Total Score data at each of the time points are included in each analysis at each time point below.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline | 122.7 (5.9) | 114.8 (16.92)
  Month 3: number analyzed (Participants) | 7 | 5
  Month 3 | 118.6 (19.11) | 117.8 (18.67)
  Month 6: number analyzed (Participants) | 6 | 3
  Month 6 | 109.4 (23.83) | 136.8 (3.43)

5. Secondary Outcome: Average LASA Overall Quality of Life at Baseline, Months 3 and 6
Description: LASA Overall Quality of Life at Baseline, Months 3 and 6. Quality of Life (QOL) was measured using the single-item Linear Analogue Self Assessment (LASA) on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The average and standard deviation of the LASA overall quality of life score are reported below at baseline, months 3 and 6.
Time Frame: Baseline to Months 3 and 6
Population: Patients who completed the LASA and had LASA Overall Quality of Life data at each of the time points are included in each analysis at each time point below.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline: number analyzed (Participants) | 6 | 7
  Baseline | 8.8 (0.75) | 6.9 (1.77)
  Month 3: number analyzed (Participants) | 7 | 5
  Month 3 | 1.0 (1.63) | 7.0 (1.22)
  Month 6: number analyzed (Participants) | 6 | 3
  Month 6 | 6.2 (3.19) | 8.7 (0.58)

6. Other Pre Specified Outcome: Correlation of Circulating Tumor Cells or Circulating Endothelial Cells Following Study Treatments With Biochemical Progression-free Survival Rate
Time Frame: 2 years
Population: Study terminated prematurely due to funding issues. Planned analysis was not performed due to the nature of the closure.
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Evaluation of Prognostic and Predictive Tissue Based Biomarkers (CTCs, CECs)
Time Frame: 2 years
Population: Study terminated prematurely due to funding issues. Planned analysis was not performed due to the nature of the closure.
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Measurements of Serum and Urine Biomarkers, and Comparison Between the Two Arms
Time Frame: 2 years
Population: Study terminated prematurely due to funding issues. Planned analysis was not performed due to the nature of the closure.
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Androgen Deprivation Therapy | No Androgen Deprivation Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androgen Deprivation Therapy (N=8) | No Androgen Deprivation Therapy (N=8)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androgen Deprivation Therapy (N=8) | No Androgen Deprivation Therapy (N=8)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 5 (12) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (17) | 1 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Taste alteration (Nervous system disorders) | 2 (3) | 1 (1)
Libido decreased (Psychiatric disorders) | 8 (26) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 7 (15) | 5 (6)
Urinary retention (Renal and urinary disorders) | 7 (13) | 5 (16)
Erectile dysfunction (Reproductive system and breast disorders) | 8 (31) | 6 (15)
Gynecomastia (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (10) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 4 (9) | 2 (2)
Flushing (Vascular disorders) | 3 (4) | 0 (0)
Hot flashes (Vascular disorders) | 7 (21) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No